CLINICAL TRIAL: NCT00222924
Title: Mitochondrial Impairment in Muscle Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 021165; R01DK049200 (NIH)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2007-12-19 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes; Obesity
Keywords: Mitochondria
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Exercise

INTERVENTIONS:
Behavioral: weight loss/ exercise

SUMMARY:
This investigation is being carried out to learn more about research findings from a study that was completed last year. Those findings revealed that within the skeletal muscle cells of individuals with type 2 diabetes, there was often damage to the mitochondria (the muscle cell's power source or the machinery of the muscle cell that produces energy). In individuals with type 2 diabetes, the liver continues to release sugar even when sugar levels are normal; the pancreas is not able to produce and release insulin normally; and the muscle and fat cells no longer respond as effectively to insulin. These defects lead to an abnormal rise of sugar in the blood. In this study, we want both to look more closely at the mitochondria and see if there is potential for improving mitochondrial functioning (improving the machinery of the muscle cell that produces energy) and reversing mitochondrial damage through a weight loss or a combined exercise/weight loss program. The program you get assigned to will be determined by a process called randomization (like a flip of a coin).

DETAILED DESCRIPTION:
Recent research from our laboratory has detected novel findings concerning damage to mitochondria within skeletal muscle in type 2 diabetes (type 2 DM), damage that is evident morphologically and by functional criteria. In this project, we propose, firstly, to more fully test this hypothesis of an impaired bio-energetic capacity, and to begin to examine the pathogenesis of damage to mitochondria in type 2 DM. We are also interested in assessing the potential for reversing damage, and improving functional capacity of mitochondria through a weight loss or a combined exercise and weight loss intervention.

The first specific aim is to measure the functional capacity of mitochondria in human skeletal muscle in type 2 DM and in those at apparent risk for type 2 DM (obese, sedentary, non-diabetic adults with the Metabolic Syndrome and/or impaired glucose tolerance). The second specific aim is to examine the morphology of mitochondria in human skeletal muscle in type 2 DM and in those at apparent risk for type 2 DM. The third specific aim is to examine the pathogenesis of mitochondrial damage in type 2 DM and in those at apparent risk for type 2 DM. The fourth specific aim is to assess whether exercise and diet can improve mitochondrial function and morphology in type 2 DM and in those at apparent risk for type 2 DM.

ELIGIBILITY:
Inclusion Criteria:

* AGE 30 to 55 years old BMI 28 to 38 kg/m2 BLOOD PRESSURE Systolic < 150 ; Diastolic < 95 SEDENTARY Currently not engaged in a regular exercise program and a VO2 max pre-training value < 55 ml/kg-fat free mass-min HEALTH (Group 1) Type 2 diabetes mellitus for < 10 years and independent in SBGM HEALTH (Group 2) Non-diabetic with impaired glucose tolerance (as per ADA) or with Metabolic Syndrome (as per NCEP-ATP III)

HEALTH Must be in good general health with no known h/o the following:

liver disease, kidney disease, PVD (including diminished pulses, or H/O thrombophlebitis), heart disease (including any h/o MI), neuromuscular disease, neurological disease (including peripheral neuropathy or muscle wasting), paresis, edema , current malignancy, or any drug or alcohol abuse, LAB VALUES Enroll if: No Proteinuria (defined as < 1+ protein on routine dipstick) Hct > 34% ALT < 80, AST < 80, Alk Phos < 240 sTSH < 8 (Group 2) 2 hr glucose on OGTT >140mg/dl but < 200mg/dl or NCEP-ATP III criteria) Triglyceride < 450 Cholesterol < 300 Negative Urine Pregnancy

Exclusion Criteria:

* (Group 1) anti-hypertensives, "statin" hypolipemics, and diabetic medications okay but exclude if taking: insulin, or a hypolipemic that is not a "statin" (Group 2) "statin" hypolipemic medications are okay. A hypolipemic that is not a "statin" will exclude.

Inability and / or unwillingness to comply with the protocol as written Previous difficulty with lidocaine or other local anesthetic Claustrophobia Wt gain or loss of > 3 kg during past 4 weeks

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49
Dates: Start 2003-12; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To measure the functional capacity of mitochondria in skeletal muscle of those with T2DM and those at increased risk of developing T2DM

SECONDARY OUTCOMES:
To assess whether exercise and diet can improve mitochondrial function and morphology.

CONTACTS AND LOCATIONS:
Overall Officials: David E. Kelley, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States